CLINICAL TRIAL: NCT01569165
Title: Effect of Water Rinsing After APF Application on Dental Plaque Acidogenicity
Brief Title: Effect of Water Rinsing After Topical Fluoride Application on Dental Plaque pH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Fatemeh Mazhari, principal investigator, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 89629
Record Dates: First submitted 2012-03-29; First posted 2012-04-03 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2012-03

CONDITIONS: Dental Caries
Keywords: Acidogenicity; Acidulated phosphate fluoride; dental plaque; water rinsing
MeSH Terms: conditions — Dental Caries; Dental Plaque

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- washing after 30 min (Experimental): washing with water after 30 min following APF treatment
  Interventions: Procedure: cleansing teeth after topical fluoride therapy
- washing after 15 min (Experimental): washing with water after 15 min following APF treatment
  Interventions: Procedure: cleansing teeth after topical fluoride therapy
- immediately washing with water (Experimental): immediately washing with water after APF treatment
  Interventions: Procedure: cleansing teeth after topical fluoride therapy
- cleansing teeth with cotton roll (Experimental): cleansing teeth with cotton roll immediately following APF treatment
  Interventions: Procedure: cleansing teeth after topical fluoride therapy
- no fluoride therapy (No Intervention): control group

INTERVENTIONS:
Procedure: cleansing teeth after topical fluoride therapy — washing with water 0, 15 or 30 min after APF treatment or cleansing teeth with cotton roll immediately following APF treatment.
  Arms: cleansing teeth with cotton roll; immediately washing with water; washing after 15 min; washing after 30 min

SUMMARY:
The aim of this study was to determine whether rinsing with water or cleansing teeth after topical fluoride therapy affect the dental plaque pH.

ELIGIBILITY:
Inclusion Criteria:

* healthy people (Without any systemic disease)
* normal unstimulated salivary rate

Exclusion Criteria:

* Active dental caries
* taking any medication with any effect on saliva rate
* taking antibiotic (or antibacterial mouth rinses) during last 4 weeks
* usig fluoride mouth rinses during last 2 weeks.

Ages: 21 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2011-02; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
dental plaque PH | the pH of 48-hour dental plaque was measured using plaque sampling method before (baseline pH) and after sucrose challenge at 5, 10,15,20,30 minutes

SECONDARY OUTCOMES:
maximum pH drop | 5,10,15,20 and 30 min after sucrose chalenge
pH recovery time | within 30 min after sucrose challenge
  time for returning to the baseline pH

CONTACTS AND LOCATIONS:
Overall Officials: fatemeh mazhari, Associate Professor, Principal Investigator — Mashhad University of Medical Siences
Locations (1):
- Dental School - Mashhad University of Medical Siences, Mashhad, Khorasan Razavi, Iran